CLINICAL TRIAL: NCT07188272
Title: Effect of High-intensity Interval Training Combined With DASH Diet on Arterial Stiffness in Hypertensive Patients: a Randomized Controlled Trial
Brief Title: Effect of High-intensity Interval Training Combined With DASH Diet on Arterial Stiffness in Hypertensive Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: September 2025
Record Dates: First submitted 2025-09-15; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Arterial Stiffness
MeSH Terms: conditions — Hypertension | interventions — Dietary Approaches To Stop Hypertension; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH diet group (Experimental): 22 patients will receive hypotensive drugs and High Intensity Interval Training ( HIIT) combined with DASH diet.
  Interventions: Dietary Supplement: DASH diet
- Comparator group (Active Comparator): 22 patients will receive hypotensive drugs and High Intensity Interval Training ( HIIT)
  Interventions: Procedure: High Intensity Interval Training

INTERVENTIONS:
Dietary Supplement: DASH diet — Eating vegetables, fruits, and whole grains Including fat-free or low-fat dairy products, fish, poultry, beans, nuts, and vegetable oils Limiting foods that are high in saturated fat, such as fatty meats, full-fat dairy products, and tropical oils such as coconut, palm kernel, and palm oils Limiting sugar-sweetened beverages and sweets
  Arms: DASH diet group
Procedure: High Intensity Interval Training — High Intensity Interval Training
  Arms: Comparator group

SUMMARY:
Cardiovascular disease (CVD) is one of the leading causes of mortality worldwide and a major risk factor for morbidity worldwide . It is necessary to reduce the incidence and risk factors of CVD, as physical activity is known to reduce mortality from CVD. Arterial stiffness and hypertension are closely related in pathophysiology. Chronic high blood pressure (BP) can lead to arterial wall damage by mechanical stress, endothelial dysfunction, increased inflammation, oxidative stress, and renin-angiotensin-aldosterone system (RAAS) activation. HIIT has been shown to be equally or even better at stimulating health benefits than moderate-intensity continuous training (MICT) and is considered a time-saving aerobic exercise for reducing arterial stiffness in HTN patients

ELIGIBILITY:
Inclusion Criteria:

* Their age< 35 up to 50 years old
* Both sexes.
* Controlled HTN ( stage 1,B.P 140-159 mmhg / 90-99 mmhg and stage 2, B.P 160-179 mmhg-100-109 mmhg )
* Hemodynamic stable. Able to provide informed consent

Exclusion Criteria:

* Uncontrolled hypertension.
* Severe HTN <180/110 mmhg
* Renal dysfunction
* Unstable cardiac conditions
* Severe pulmonary disease that limit exercise
* Impaired cognition
* Musculoskeletal problems that made it difficult to do exercise

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Velocity | each week
  normal level 60-100 per minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Waleed Mohamed Abdelmohsen Abdelsalalm, Minya, Egypt